CLINICAL TRIAL: NCT00855894
Title: An Open-label Phase II Multicenter Study of the Safety and Activity (as Measured by FDG-PET Imaging Changes) of the Combination of Erlotinib and Pertuzumab in Patients With Relapsed Non-small Cell Lung Cancer
Brief Title: A Study of the Combination of Erlotinib and Pertuzumab in Patients With Relapsed Non-small Cell Lung Cancer
Acronym: PENGUIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOC4603g; GO01357 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Tarceva; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pertuzumab; Erlotinib Hydrochloride

ARMS (1):
- Pertuzumab + erlotinib (Experimental): Patients received pertuzumab 840 mg intravenously (IV) 1 time (loading dose) followed by 420 mg IV (maintenance dose) every 3 weeks (q3w) plus erlotinib 150 mg orally once a day which was reduced to 100 mg orally once a day in a protocol amendment dated 19 May 2010.
  Interventions: Drug: Pertuzumab; Drug: Erlotinib

INTERVENTIONS:
Drug: Pertuzumab — After a single administration of a loading dose of 840 mg IV, patients received a maintenance dose of 420 mg IV every 3 weeks (q3w).
  Other Names: Perjeta
Drug: Erlotinib — Patients received 150 mg orally once a day which was reduced to 100 mg orally once a day in a protocol amendment dated 19 May 2010.
  Other Names: Tarceva

SUMMARY:
This was a Phase II, open-label, single-arm, single-stage, multicenter trial in patients with relapsed non-small cell lung cancer (NSCLC), with the objective of assessing the activity of the combination of erlotinib and pertuzumab on the basis of the endpoint of FDG-PET response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC).
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Recurrent or progressive disease after receiving at least 1, but no more than two, chemotherapy regimens for advanced or metastatic NSCLC.
* Recovery from reversible acute effects of prior anti-cancer therapy (chemotherapy, radiotherapy, or investigational treatment) to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade ≤ 1 (excluding alopecia).
* Ability to comply with the study and follow-up procedures, including all specified imaging studies.
* Ability to take oral medication.
* Life expectancy ≥ 3 months.
* Measurable disease on computed tomography (CT).
* At least 1 extracerebral lesion on 2-deoxy-2-[18F]fluoro-D-glucose-positron emission tomography (FDG-PET) scan that is suitable for response assessment, that is measurable, and ≥ 15 mm on CT.
* Left ventricular ejection fraction (LVEF) ≥ 50%, as determined by echocardiogram or MUltiple Gated Acquisition (MUGA) scan.
* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the patient and/or partner.
* Availability and willingness to provide sufficient tumor tissue for testing for epidermal growth factor receptor (EGFR) mutations, and other human epidermal growth factor receptor (HER) pathway and NSCLC-related biomarkers.

Exclusion Criteria:

* Prior treatment with an investigational or marketed agent for the purpose of inhibiting HER family members (including HER1, HER2, HER3, and HER4). This includes, but is not limited to erlotinib, gefitinib, pertuzumab, cetuximab, and panitumumab.
* Chemotherapy, radiotherapy, or investigational treatment within 28 days of start of study (ie, prior to Day 0) or from which patients have not yet recovered.
* Inability to take oral medications, disease affecting gastrointestinal absorption, or prior surgical procedure affecting gastrointestinal absorption.
* Uncontrolled diabetes.
* Clinical or radiographic evidence of new or progression of pre-existing central nervous system (CNS) metastases.
* Current severe, uncontrolled systemic disease (eg, clinically significant cardiovascular, pulmonary, or metabolic disease; wound-healing disorders; ulcers; or bone fractures).
* Current uncontrolled hypertension or unstable angina.
* History of congestive heart failure (CHF) of any New York Heart Association (NYHA) criteria, or serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia).
* History of myocardial infarction within 6 months of enrollment or history of unstable angina.
* Any evidence of an unstable infection as suggested by an infectious process, coupled with hypotension and/or tachycardia and/or fever and/or positive blood culture.
* Known human immunodeficiency virus (HIV) infection.
* Uncontrolled hypercalcemia.
* Pregnancy or lactation.
* History of another malignancy in the past 2 years, unless the malignancy has been adequately treated, is currently not detectable, and is associated with a 5-year survival > 90%.
* Claustrophobia.
* Any other disease, condition, physical examination finding, or clinical laboratory finding that, in the opinion of the investigator, makes the patient inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pirzkall, M.D., Study Director — Genentech, Inc.
Locations (10):
- United States (4):
  - Los Angeles, California
  - Rancho Mirage, California
  - Omaha, Nebraska
  - Seattle, Washington
- Australia (6):
  - Adelaide
  - Chermside
  - East Melbourne
  - Heidelberg
  - Herston
  - Sydney

REFERENCES:
- [Derived] Hughes B, Mileshkin L, Townley P, Gitlitz B, Eaton K, Mitchell P, Hicks R, Wood K, Amler L, Fine BM, Loecke D, Pirzkall A. Pertuzumab and erlotinib in patients with relapsed non-small cell lung cancer: a phase II study using 18F-fluorodeoxyglucose positron emission tomography/computed tomography imaging. Oncologist. 2014 Feb;19(2):175-6. doi: 10.1634/theoncologist.2013-0026. Epub 2014 Jan 23. PMID 24457379

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were considered to have completed the study if they were alive at their last survival follow-up visit prior to 10 Nov 2011, which was 1 year after the last patient was enrolled, or they were continuing treatment per Amendment 3 of the study protocol (1 patient).
Period: Overall Study
Arm/Group | Pertuzumab + Erlotinib
Started | 41
Completed | 8
Not Completed | 33
Not completed — Death | 31
Not completed — Patient's decision | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 60.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a 2-deoxy-2-[18F]Fluoro-D-glucose-positron Emission Tomography (FDG-PET) Response at Day 56 in All Patients and in Epidermal Growth Factor Receptor (EGFR) Mutant and Wild-type Subgroups
Description: The assessment of FDG-PET response was performed by a central reading site. PET response was based on the maximum standard uptake value (SUVmax) of up to 5 regions of interest (ROI). The tumor ROIs were identified for each patient on pretreatment FDG-PET scans and corresponded to a subset of the target lesions identified for Response Evaluation Criteria for Solid Tumors (RECIST) analysis. Specifically, the SUVmax of each ROI on the on-treatment scans was compared with the SUVmax on the corresponding pretreatment scan and the percent change was calculated. When there was more than 1 ROI, the overall percent change in SUVmax was the arithmetic mean of the percent changes in SUVmax for each of the ROIs (mSUVmax). An PET response is defined as a decrease of ≥ 20% in mSUVmax. EGFR mutation status was assessed in tumor tissue samples taken from each patient.
Time Frame: Baseline to Day 56
Population: All 41 patients treated with pertuzumab and erlotinib were evaluable for analysis. Patients with a missing Day 56 assessment were deemed non-responders. Tumor tissue samples were only available for 32 patients for EGFR mutation status analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 41
Percentage of patients
  In all patients | 19.5 [9.2 to 33.9]
  In patients with EGFR mutation(s), n=9 | 66.7 [29.9 to 90.2]
  In patients with wild-type EGFR, n=23 | 8.7 [1.6 to 26.8]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dosing with pertuzumab and erlotinib to the first occurrence of disease progression (PD), as determined by the investigator and based on computed tomography using Response Evaluation Criteria in Solid Tumors (RECIST), or death from any cause, whichever comes first. PD was defined as ≥ 20% increase in the sum of the longest diameter of target lesions (TL), taking as reference the smallest sum longest diameter recorded since treatment started, the unequivocal progression of existing non-target lesions (non-TL), or the appearance of 1 or more new lesions. TLs were selected on the basis of their size (those with the longest diameter) and their suitability for accurate repeated measurements by imaging techniques or clinically. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, were identified as TLs. All other lesions (or sites of disease) were identified as non-TLs.
Time Frame: Baseline to the end of the study (up to 3 years)
Population: All 41 patients treated with erlotinib and pertuzumab. Patients who had not progressed or died at the time of analysis for PFS were censored at the date of their last tumor assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 41
Months | 1.9 [1.87 to 3.38]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of first dosing with pertuzumab and erlotinib until the date of patient death from any cause.
Time Frame: Baseline to the end of the study (up to 3 years)
Population: All 41 patients treated with erlotinib and pertuzumab. Patients who had not died at the time of analysis for OS were censored at the date of last contact.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 41
Months | 8.7 [4.70 to 9.99]

4. Secondary Outcome: Percentage of Patients With an Objective Response (OR)
Description: OR was defined as a complete response (CR) or a partial response (PR) as determined by the investigator and based on computed tomography (CT) using Response Evaluation Criteria in Solid Tumors (RECIST) on 2 consecutive occasions at least 4 weeks apart. A complete response was defined as the disappearance of all target and non-target lesions and normalization of tumor marker level. A partial response was defined as ≥ 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter, or the persistence of 1 or more non-target lesions and/or the maintenance of a tumor marker level above the normal limits.
Time Frame: Baseline to the end of the study (up to 3 years)
Population: All 41 patients treated with erlotinib and pertuzumab.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 41
Percentage of patients | 7.3 [2.0 to 19.0]

5. Secondary Outcome: Percentage of Patients With Disease Control (DC) at Day 56
Description: DC was defined as a CR, a PR, or stable disease (SD) as determined by the investigator and based on CT using RECIST. A CR was defined as the disappearance of all target (TL) and non-target lesions (nTL). A PR was defined as ≥ 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline sum longest diameter, or the persistence of 1 or more nTLs and/or maintenance of a tumor marker level (TML) above normal limits. For TLs, SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter (SSLD) since treatment started. For nTLs, SD was defined as the persistence of 1 or more lesions and/or maintenance of a TML above normal limits. PD was defined as ≥ 20% increase in the SLD of TLs, taking as reference the SSLD recorded since treatment started, the appearance of 1 or more new lesions, or the unequivocal progression of existing nTLs.
Time Frame: Baseline to Day 56
Population: All 41 patients treated with erlotinib and pertuzumab.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Pertuzumab + Erlotinib
Number analyzed (Participants) | 41
Percentage of patients | 31.7 [19.0 to 46.9]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were reported from the time of enrollment in the study up to 30 days after the last day of treatment or study discontinuation, whichever was later (up to 3 years).
Description: Adverse events are reported for all patients who received at least 1 dose of study treatment.
Arm/Group | Pertuzumab + Erlotinib
Serious Adverse Events (participants affected / at risk) | 18/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab + Erlotinib (N=41)
Anaemia (Blood and lymphatic system disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Pneumatosis intestinalis (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Infection (Infections and infestations) | 1
Pharyngeal abscess (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Tumor invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab + Erlotinib (N=41)
Anaemia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 3
Dry eye (Eye disorders) | 7
Conjunctivitis (Eye disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 36
Nausea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 21
Stomatitis (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 28
Mucosal infalmmation (General disorders) | 22
Oedema peripheral (General disorders) | 5
Chest pain (General disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Paronychia (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 3
Weight decreased (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 26
Hypokalaemia (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Hypoalbumaemia (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 9
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 26
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash generalised (Skin and subcutaneous tissue disorders) | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.